CLINICAL TRIAL: NCT05551143
Title: R2P Field Test of the EMS LiftKit: Validating Usability, Usefulness, Desirability, and Effects on Musculoskeletal Injuries in EMS Providers Working in Urban, Suburban, and Rural Communities
Brief Title: R2P Field Test of the EMS LiftKit: Validating Usability, Usefulness, Desirability, and Effects on Musculoskeletal Injuries in EMS Providers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Steve Lavender, Associate Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LiftKit
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Musculoskeletal Disorder
Keywords: EMS; Ergonomics; Musculoskeletal Disorders; Back Injury; Firefighter
MeSH Terms: conditions — Musculoskeletal Diseases; Back Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LiftKit Intervention (Experimental): All participants will have access to the LiftKit that provides them with a set of tools that should reduce the physical demands experienced by EMS providers when lifting and moving patients in their homes, thereby reducing the risk of musculoskeletal disorders (MSDs).
  Interventions: Other: LiftKit

INTERVENTIONS:
Other: LiftKit — The LiftKit contains 7 tools that could assist EMS providers when lifting/moving patients. These tools are:
  1. Simple Strap - A sling to lift a seated patient
  2. Strap and slide stick - A strap system for raising a supine patient to a sitting posture.
  3. Slip Preventer- An envelope that goes over the patients feet with high friction straps for the EMS providers to stand on that prevent the patient from sliding forward when lifted.
  4. Drag Straps - straps with handles that can be clipped on tarps used to drag patients
  5. The Binder Lift - a vest with handles that allow EMS providers to easily get hold of patient they need to lift.
  6. Patient Turning Straps - a way to log-roll a patient that in on the floor while in a standing posture.
  7. The ELK - an inflatable seat cushion that can raise a patient who in the floor to chair level

SUMMARY:
The long-term goal of our research program is to reduce the high incidence of musculoskeletal injury associated with person-handling tasks performed by EMS providers/responders (NORA Public Safety Industry Sector). The literature shows the significant burden of these injuries, many of which affect the back and are debilitating. There is a need for effective ergonomic tools that can assist EMS providers in the patient handling tasks encountered in patient homes, particularly those patient handling situations that include restricted or tight spaces. To address this need, our prior work identified a set of potential ergonomic solutions, using a participatory process with EMS providers, for physically challenging and frequently occurring patient handling tasks that occur in patient homes. A final product of this prior work was the development of the LiftKit, which is a collection of seven tools that were shown in biomechanical validation studies with EMS providers to effectively reduce physical demands during simulated patient handling tasks in a laboratory setting. The overall objective of this proposed research-to-practice application is to evaluate the LiftKit's seven patient handling tools (interventions) in the field to assess their usability, usefulness, and desirability, as well as their impact with regards to preventing musculoskeletal injuries incurred during EMS patient handling tasks. In this field study, 30 LiftKits will be placed on EMS vehicles that service urban, suburban, and rural communities. Given the three-shift operation used by fire-service based EMS departments, there is the potential to recruit between 180 and 270 EMS providers for the study. Immediately following the training on how to use the tools and at 4, 8, and 12 months following the training, participants will be interviewed and questioned about each tools' usability, usefulness, and desirability. Frequency of each tool's use will be assessed with a questionnaire at the time of the interview and a daily Run-Use survey tool. Musculoskeletal injury data due to patient handling tasks during the 12 month follow-up period will be compared with injury data from the three-year period prior to study initiation. The final product of this work will provide the important evidence needed to widely promote the adoption of the ergonomic tools within the LiftKit, in order to reduce MSD injury risk to EMS providers associated with common patient handling tasks.

ELIGIBILITY:
Inclusion Criteria:

* Working EMS providers

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Reported Musculoskeletal Injuries | 12 months
  Injuries that are due to patient handling tasks within the patient's home.

SECONDARY OUTCOMES:
Usability, Usefulness, and Desirability of the tools within the LiftKit | 12 months
  Survey assessments

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No